CLINICAL TRIAL: NCT02968992
Title: Effects of Lactoferrin on Chronic Inflammation in the Elderly
Brief Title: Effects of rhLactoferrin on Chronic Inflammation in the Elderly
Acronym: ELCIE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Ventria Bioscience (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00094982; R21AG053681-01 (NIH)
Record Dates: First submitted 2016-11-15; First posted 2016-11-21 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Inflammation; Cognitive Deterioration
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: •Randomized: Participants are assigned to intervention groups by chance
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- rhLactoferrin (Experimental): rH lactoferrin will be provided by Ventria Biosciences. Each capsule will contain 250 mg of rH lactoferrin as active ingredient. Subjects will receive 1500 mg of lactoferrin in capsule form twice a day. Dosing will be six 250 mg capsules twice a day for six months.
  Interventions: Drug: rhLactoferrin
- Placebo (Placebo Comparator): Matching placebo capsule will be provided by Ventria Biosciences and six capsules twice a day will be provided to the subjects in this arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: rhLactoferrin — Eligible participants will be provided with Recombinant Human lactoferrin (rhLF) in 250 mg capsules along with detailed instructions for taking the study drug and they will be asked to take six 250 mg capsules twice a day and to keep a daily dosing dairy.
  Arms: rhLactoferrin
Other: Placebo — Eligible participant will be provided with placebo in capsules of 250 mg along with detailed instructions for taking the placebo. Participants will be asked to take six 250 mg capsules twice a day and to keep a daily dosing dairy.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate how recombinant human lactoferrin (rhLF) which is a partially iron saturated form of lactoferrin produced and purified from rice grain may improve mobility and memory in older adults with chronic inflammation. Lactoferrin, is a known multifunctional protein, and has been shown to have anti-inflammatory effects. A recombinant human version of this protein was recently developed and produced from rice. This is now available from the Ventria Bioscience Company in a controlled, pharmaceutical grade capsule. As part of this double blinded and randomized study, participants will take daily dosages of recombinant human lactoferrin (rhLF) or its matched placebo; to measure the effects of rhlactoferrin on chronic inflammation and its association with improving mobility and memory over a 6 month time period. During the study all participants will be asked to provide blood samples and will have physical and cognitive tests administered to them. By measuring biomarkers in the blood as well as changes in physical and cognitive measures, the investigators will gain an understanding of how rhlactoferrin may safely improve measures of chronic inflammation in older adults. As well as a better understanding of whether it has the potential to meaningfully influence important measures of physical and cognitive function known to be influenced by Chronic Inflammation (CI).

DETAILED DESCRIPTION:
The primary objective of this study is to examine in a double blinded and randomized trial the efficacy of Recombinant Human lactoferrin (rhLF) in reducing chronic inflammation as measured by IL-6 and sTNFR1 in the bloodstream. The primary end point is to gather information about the tolerability of and adherence to oral rhlactoferrin (rhLF) among older adults with CI over a six-month period. The exploratory objective is to assess the efficacy of rhlactoferrin (rhLF) in attenuating cognitive decline as measured by the Digit Symbol Substitution Test and Trail Making Test, as well as improving physical mobility as measured by performance on 4 meter and six-minute walk tests. Further physical and functional measurement data will be gather using an Acti-graph link Activity monitor, the raw data collected will be used to : (i) characterize cumulative daily activity, (ii) assess daily circadian patterns of activity, (iii) assess physical activity variability, (iv) model patterns of daily activity, and (iv) estimate walking speed. This additional data will complement mobility measures by describing function enacted in daily life

ELIGIBILITY:
Inclusion Criteria:

* Age 70 and older
* able to complete 4- meter timed walk; walking speed <1.0 m/sec
* serum IL-6 level ≥ 2.5 pg/ml or TNFR1 level ≥1500 pg/ml

Exclusion Criteria:

* Daily anti-inflammatory drug use (prednisone, Advil, Aleve, Remicade, Enbrel, methotrexate, standing nonsteroidal anti-inflammatory drugs (NSAID), aspirin greater than 325 mg per day)
* lower extremity mobility disability caused by Parkinson's disease,
* cerebral vascular accident (CVA) with residual motor deficit,
* severe osteoarthritis or rheumatoid arthritis
* symptomatic claudication
* hospitalization within 3 months for myocardial infarction (MI), angina, infection requiring antibiotics, or joint replacement.
* Mini-Mental State Examination (MMSE) < 21.
* Lactose intolerant
* allergy or intolerance to bovine products
* being a vegan (since vegans will want to avoid Bovine products.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerermy D. Walston, MD, Principal Investigator — Johns Hopkins Universtiy
Locations (1):
- Jeremy D. Walston, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | rhLactoferrin | Placebo
Started | 18 | 18
Completed | 18 | 17
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rhLactoferrin | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.6 (6.6) | 79.6 (5.6) | 81.1 (6.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 17 | 34
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 14 | 15 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Count of Participants; unit: Participants]
  BMI ≥ 30 | 5 | 8 | 13
  BMI < 30 | 13 | 10 | 23
Physical mobility as measured by 4 meter walk test [Mean (Standard Deviation); unit: m/sec] — A standard measurement of 4 meters is marked on a flat, long floor surface. The test taker is asked to walk the length at their usual pace while the test giver is recording the time with a stop watch. This test is repeated twice, and the average of the two recorded times is used as the data point. Population: A total of 36 participants entered the study. One participant in the placebo group later dropped out and therefore was not included in the analysis.
  m/sec
    number analyzed (Participants) | 18 | 17 | 35
    (all) | 0.78 (0.17) | 0.78 (0.13) | 0.78 (0.15)
Physical strength as measured by grip strength [Mean (Standard Deviation); unit: kg] — Hand grip strength is measured by the amount of static force that the hand can squeeze around a dynamometer. An administrator recorded the reading on the device. The force was measured in kilograms. Population: A total of 36 participants entered the study. One participant in the placebo group later dropped out and therefore was not included in the analysis.
  kg
    number analyzed (Participants) | 18 | 17 | 35
    (all) | 26.2 (7.3) | 25.3 (6.7) | 25.8 (6.9)
Physical mobility as measured by 6 minute walk test [Mean (Standard Deviation); unit: meters] — A measured course is set up in an open area on a hard flat surface. The test taker walks on this measured course for 6 minutes, and the test administrators calculates the distance traveled over 6 minutes. The test taker is allowed to rest as is needed. Population: A total of 36 participants entered the study. One participant in the placebo group later dropped out and therefore was not included in the analysis. One participant in the treatment group declined to complete the test.
  meters
    number analyzed (Participants) | 17 | 17 | 34
    (all) | 358.9 (124.3) | 345.8 (88.9) | 352.3 (106.6)
Log Total Activity Count [Mean (Standard Deviation); unit: Log Total Activity Count] — Log total activity count was determined using the Acti-Graph® Link Activity monitor which generates a comprehensive assessment of daily free-living activity. Participants wore the monitor for 7 days. Activity counts are proprietary units generated by the Actigraph company software, Actilife. Counts are unitless quantities of physical activity compiled into one-minute intervals across three planes of movement. The vector magnitude of the sum of square of these counts generate the total activity per minute, per hour and per day. Population: A total of 36 participants entered the study, one participant in the placebo group later dropped out and therefore was not included in the analysis.
  Log Total Activity Count
    number analyzed (Participants) | 18 | 17 | 35
    (all) | 14.26 (0.35) | 14.46 (0.28) | 14.35 (0.33)
Attenuating cognitive decline as measured by the trail making test A and B [Mean (Standard Deviation); unit: seconds] — For test A, the individual is given a sheet of paper that has the numbers 1-25 within individual circles randomly distributed. The individual is asked to connect the numbers sequentially. The score is recorded as the time it takes to complete the task in seconds. For test B, the individual is given a piece of paper that has numbers 1-13 and letters A-L. Each letter or number is inside of a circle. The test taker is instructed to draw a line from one number to the next letter (ie. 1 to A to 2 to B etc.). The score is the seconds it takes to complete the task. Population: A total of 36 participants entered the study. One participant in the placebo group later dropped out and therefore was not included in the analysis of test A and test B data. One additional participant in the placebo group was unable to complete Trail Making Test B, so they were not included in the analysis.
  seconds
    Test A: number analyzed (Participants) | 18 | 17 | 35
    Test A | 48.3 (16.7) | 54.1 (28.9) | 51.1 (23.3)
    Test B: number analyzed (Participants) | 18 | 16 | 34
    Test B | 101.1 (34.6) | 109.3 (49.3) | 104.9 (41.7)
Attenuating cognitive decline as measured by the digital symbol substitution test [Mean (Standard Deviation); unit: Correct answers] — The test taker is given a key consisting of numbers 1-9 that are paired with a unique symbol. Below the key is a randomly generated list of the numbers repeated several times. The test taker is allowed 90 seconds to assign the correct symbol to the number on the list. The test administrator then scores the number of correct answers over the 90 second test time, and assigns a total score based on one point for each correct answer. Population: A total of 36 participants entered the study. One participant in the placebo group later dropped out and therefore was not included in the analysis.
  Correct answers
    number analyzed (Participants) | 18 | 17 | 35
    (all) | 33 (12) | 31 (10) | 32 (11)

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Rhlactoferrin on Serum Levels of Interleukin-6 (IL-6)
Description: The effect of rhlactoferrin on serum levels (picogram/milliliter) of Interleukin-6 (IL-6) will be assessed as a measure of the percentage change of IL-6 serum levels from baseline
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: Percent change of IL-6
Arm/Group | rhLactoferrin | Placebo
Number analyzed (Participants) | 18 | 17
Percent change of IL-6 | -0.640 (1.137) | 0.932 (0.265)

2. Primary Outcome: The Effect of Rhlactoferrin on Serum Levels of Tumor Necrosis Factor Alpha Receptor 1 (TNFR1)
Description: The effect of rhlactoferrin on serum levels (picogram/milliliter) of tumor necrosis factor alpha receptor 1 (TNFR1) assessed as a measure of the percentage change of serum TNFR1 levels from baseline
Time Frame: From baseline to 6 months
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | rhLactoferrin | Placebo
Number analyzed (Participants) | 18 | 17
Percent change from baseline | 19.709 (85.084) | 140.748 (43.24)

3. Secondary Outcome: Attenuating Cognitive Decline as Measured by the Digital Symbol Substitution Test
Description: The test taker is given a key consisting of numbers 1-9 that are paired with a unique symbol. The test taker is allowed 90 seconds to assign the correct symbol to the number on the list. The test administrator then scores the number of correct answers over the 90 second test time, and assigns a total score based on one point for each correct answer and therefore a higher score is a better outcome.
Time Frame: At 6 months
Measure: Mean (95% Confidence Interval); unit: correct responses
Arm/Group | rhLactoferrin | Placebo
Number analyzed (Participants) | 18 | 17
correct responses | 31.61 [26.07 to 37.16] | 31 [25.42 to 36.58]

4. Secondary Outcome: Attenuating Cognitive Decline as Measured by the Trail Making Test A and B.
Description: For test A, the test taker is given a sheet of paper that has the numbers 1-25 within individual circles randomly distributed on the page. The test taker is asked to connect the numbers sequentially over a period of 4 minutes (240 seconds). The score is recorded as the time it takes to complete the task in seconds. For test B, the test taker is given a piece of paper that has numbers 1-13 and letters A-L. Each letter or number is inside of a circle. The test taker must then draw a line from one circled number to the next circled letter (ie. 1 to A to 2 to B to 3 to C etc.) over a period of 6 minutes (360 seconds). The time it takes to complete this task is recorded in seconds.
Time Frame: At 6 months
Population: A total of 36 participants entered the study. One participant in the placebo group later dropped out and therefore was not included in the analysis. One additional participant in the placebo group was unable to complete Trail Making Test B, so they were not included in the analysis.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | rhLactoferrin | Placebo
Number analyzed (Participants) | 18 | 17
seconds
  Trail Making Test A | 33.11 [26.36 to 39.85] | 42.68 [35.89 to 49.47]
  Trail Making Test B: number analyzed (Participants) | 18 | 16
  Trail Making Test B | 122.73 [92.31 to 153.14] | 131.24 [100.61 to 161.87]

5. Secondary Outcome: Physical Mobility as Measured by 4 Meter Walk Test
Description: A standard measurement of 4 meters is marked on a flat, long floor surface. The test taker is asked to walk the length at their usual pace while the test giver is recording the time with a stop watch. This test is repeated twice, and the average of the two recorded times is used as the data point.
Time Frame: At 6 months
Measure: Mean (95% Confidence Interval); unit: m/sec
Arm/Group | rhLactoferrin | Placebo
Number analyzed (Participants) | 18 | 17
m/sec | 0.786 [0.701 to 0.871] | 0.767 [0.681 to 0.852]

6. Secondary Outcome: Physical Mobility as Measured by 6 Minute Walk Test
Description: A measured course is set up in an open area on a hard flat surface. The test taker walks on this measured course for 6 minutes, and the test administrators calculates the distance traveled over 6 minutes. The test taker is allowed to rest as is needed.
Time Frame: At 6 months
Measure: Mean (95% Confidence Interval); unit: meter
Arm/Group | rhLactoferrin | Placebo
Number analyzed (Participants) | 18 | 17
meter | 359.66 [303.02 to 416.3] | 334.94 [279.48 to 390.4]

7. Secondary Outcome: Tolerability of Oral rhLactoferrin as Assessed by Patient Diary of Total Number of Side Effects
Description: Study coordinators administered side effect questionnaire at each visit and via phone every two weeks during the treatment period.
Time Frame: From baseline through 6 months.
Measure: Mean (Standard Deviation); unit: Side effects/100 treatment days
Arm/Group | rhLactoferrin | Placebo
Number analyzed (Participants) | 18 | 17
Side effects/100 treatment days | 2.23 (3.16) | 4.77 (4.23)

8. Secondary Outcome: Physical Strength as Measured by Grip Strength
Description: Hand grip strength is measured by the amount of static force that the hand can squeeze around a dynamometer. An administrator recorded the reading on the device. The force was measured in kilograms.
Time Frame: At 6 months
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | rhLactoferrin | Placebo
Number analyzed (Participants) | 18 | 17
kg | 23.493 [20.694 to 26.337] | 20.294 [17.34 to 23.157]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | rhLactoferrin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/18
Other Adverse Events (participants affected / at risk) | 13/18 | 15/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhLactoferrin (N=18) | Placebo (N=18)
Hospitalization (Infections and infestations) | 0 (0) | 1 (1) — Participant suffered an infection from cat bite, which required hospitalization, and he was withdrawn from study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rhLactoferrin (N=18) | Placebo (N=18)
Diarrhea (Gastrointestinal disorders) | 2 | 5
Skin rash (Skin and subcutaneous tissue disorders) | 0 | 1
Loss of Appetite (General disorders) | 2 | 1
Fatigue (General disorders) | 5 | 4
Fever/chills (General disorders) | 4 | 0 — Fever or chills were associated with respiratory infections
Constipation (Gastrointestinal disorders) | 3 | 4
Other conditions (General disorders) | 12 | 9 — Other conditions consist of any other medical issues that were not included in the standard side effects.

LIMITATIONS AND CAVEATS:
The primary limitation of this study was the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT02968992/Prot_SAP_001.pdf